CLINICAL TRIAL: NCT03673397
Title: The Acute Effect of Aerobic Exercise on Sleep in Patients With Depression: a Randomized Controlled Trial
Brief Title: The Acute Effect of Aerobic Exercise on Sleep in Patients With Depression
Acronym: EASED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oberwaid AG (Other)
Collaborators: Institute for Exercise and Health Sciences, University of Basle, Switzerland (Other); University of Zurich (Other); University of Basel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EASED-trial
Record Dates: First submitted 2018-06-28; First posted 2018-09-17 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Depression; Sleep; Sleep Disorder; Sleep Disturbance; Sleep Fragmentation; Sleep Initiation and Maintenance Disorders; Insomnia; Insomnia, Psychophysiological; Insomnia Due to Other Mental Disorder; Insomnia Related to Another Mental Condition
Keywords: Exercise; Sleep; Depression; Heart rate variability; Blood pressure; randomized controlled trial; polysomnography
MeSH Terms: conditions — Depression; Sleep Wake Disorders; Parasomnias; Sleep Deprivation; Sleep Initiation and Maintenance Disorders; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise (Experimental): Patients allocated to the intervention group will perform a single bout of supervised aerobic exercise. The starting time will be approximately 1630 hrs. The exercise mode will be a bicycle ergometer. After a warm-up period, during which the intensity is gradually increased, an intensity of 80% of the individual anaerobic threshold will be maintained for 30 minutes. The intensity level was chosen based on clinical experience that this corresponds to an approximate rate of perceived exertion of 13 (on a scale from 6-20) in this population.
  Interventions: Behavioral: Aerobic exercise, bicycle ergometer
- Control (No Intervention): Individuals allocated to the control group will be placed in a room with analogous conditions to the exercise group concerning light, temperature and absence of music at the same time as individuals performing the exercise intervention. The control group will be asked to remain seated and read magazines.

INTERVENTIONS:
Behavioral: Aerobic exercise, bicycle ergometer — Exercise performed below individual anaerobic threshold for 30 minutes
  Arms: Aerobic exercise

SUMMARY:
The aim of this trial is to investigate the effects of a single bout of aerobic exercise on sleep in patients with depression.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

The primary objective of this study is to evaluate whether a single bout of aerobic exercise improves sleep efficiency more than a control condition in patients with depression.

SECONDARY OBJECTIVES:

Secondary objectives are to assess the effects of a single bout of aerobic exercise on 1) sleep continuity, 2) sleep architecture, 3) pre-sleep arousal, 4) subjective sleep quality, 5) daytime sleepiness, 6) nocturnal blood pressure, 7) heart rate variability, and 8) the frequency and severity of adverse events.

DESIGN:

This will be a two-arm parallel group, randomized, outcome assessor blinded, controlled, superiority trial. According to sample size calculation a total of 92 patients will be randomized using minimization. The trial will take place in the first five days of the patients' psychosomatic in-patient rehabilitation in the clinic OBERWAID, St.Gallen, Switzerland. The study visits are scheduled is as follows:

Day 0-2: Screening, inclusion, and graded exercise test to determine exercise intensity of intervention

Day 3: Questionnaires for background information

Night 1 (day 3-4): Baseline polysomnography and sleep related questionnaires

Day 4: Randomized allocation (control or exercise condition) and performing corresponding intervention

Night 2 (day 4-5): Follow-up polysomnography and sleep related questionnaires

Day 5: Daytime sleepiness questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Inpatient psychosomatic rehabilitation in the clinic OBERWAID, St.Gallen, Switzerland
* Age: ≥18 and ≤65 years old
* Primary diagnosis of depression (F32, F33) without psychotic episode according to International Statistical Classification of Diseases, 10th edition

Exclusion Criteria:

* Regular use of hypnotic agents (patients were included if no hypnotic agents were taken 2 weeks prior to study participation)
* Factors precluding exercise testing or training
* Use of beta-blockers (with the exception of Carvedilol & Nebivolol)
* Use of opioids
* History of epilepsy
* Restless legs syndrome defined by ≥7 points on the restless legs syndrome screening questionnaire (RLSSQ)
* Moderate or severe sleep apnea defined by an oxygen desaturation index (ODI) ≥15 in the first polysomnography.
* Morbid adiposity with BMI >40

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in sleep efficiency (%) at follow-up assessed by polysomnography | Baseline (night 1) and follow-up (night 2)
  Calculated as (total sleep time / total recording time) * 100. Higher values represent a better outcome. A one-way ANCOVA will be computed with baseline sleep efficiency (%) and minimization factors as covariates, intervention as the independent variable, and follow-up sleep efficiency (%) as the dependent variable.

SECONDARY OUTCOMES:
Change from baseline in wake after sleep onset (minutes) at follow-up assessed by polysomnography | Baseline (night 1) and follow-up (night 2)
  Calculated as time awake after first sleep episode. Lower values represent better outcome. A one-way ANCOVA will be computed with baseline wake after sleep onset and minimization factors as covariates, intervention as the independent variable, and follow-up wake after sleep onset as dependent variables.
Change from baseline in sleep onset latency (minutes) at follow-up assessed by polysomnography | Baseline (night 1) and follow-up (night 2)
  Calculated as time between lights-off marker and first epoch of any sleep stage. Lower values represent better outcome. A one-way ANCOVA will be computed with baseline sleep onset latency and minimization factors as covariates, intervention as the independent variable, and follow-up sleep onset latency as dependent variables.
Change from baseline in number of awakenings at follow-up assessed by polysomnography | Baseline (night 1) and follow-up (night 2)
  Calculated as number of wake periods of at least two epochs after sleep onset. Lower values represent better outcome. A one-way ANCOVA will be computed with baseline number of awakenings and minimization factors as covariates, intervention as the independent variable, and follow-up number of awakenings as dependent variables.
Change from baseline in stage 1 sleep (% of total sleep time and minutes) at follow-up assessed by polysomnography | Baseline (night 1) and follow-up (night 2)
  Calculated as Stage 1 sleep (in minutes and % of total sleep time). A one-way ANCOVA will be computed with baseline stage 1 sleep (% of total sleep time and minutes) and minimization factors as covariates, intervention as the independent variable, and follow-up stage 1 sleep (% of total sleep time and minutes) as dependent variables.
Change from baseline in stage 2 sleep (% of total sleep time and minutes) at follow-up assessed by polysomnography | Baseline (night 1) and follow-up (night 2)
  Calculated as Stage 2 sleep (in minutes and % of total sleep time). A one-way ANCOVA will be computed with baseline stage 2 sleep (% of total sleep time and minutes) and minimization factors as covariates, intervention as the independent variable, and follow-up stage 2 sleep (% of total sleep time and minutes) as dependent variables.
Change from baseline in stage 3 sleep (% of total sleep time and minutes) at follow-up assessed by polysomnography | Baseline (night 1) and follow-up (night 2)
  Calculated as Stage 3 sleep (in minutes and % of total sleep time). A one-way ANCOVA will be computed with baseline stage 3 sleep (% of total sleep time and minutes) and minimization factors as covariates, intervention as the independent variable, and follow-up stage 3 sleep (% of total sleep time and minutes) as dependent variables.
Change from baseline in rapid eye movement sleep (% of total sleep time and minutes) at follow-up assessed by polysomnography | Baseline (night 1) and follow-up (night 2)
  Calculated as rapid eye movement sleep (in minutes and % of total sleep time). A one-way ANCOVA will be computed with baseline rapid eye movement sleep (% of total sleep time and minutes) and minimization factors as covariates, intervention as the independent variable, and follow-up rapid eye movement sleep (% of total sleep time and minutes) as dependent variables.
Change from baseline in light sleep (% of total sleep time and minutes) at follow-up assessed by polysomnography | Baseline (night 1) and follow-up (night 2)
  Calculated as sum of Stage 1 & 2 sleep (in minutes and % of total sleep time). A one-way ANCOVA will be computed with baseline light sleep (% of total sleep time and minutes) and minimization factors as covariates, intervention as the independent variable, and follow-up light sleep (% of total sleep time and minutes) as dependent variables.
Change from baseline in non-rapid eye movement sleep (% of total sleep time and minutes) at follow-up assessed by polysomnography | Baseline (night 1) and follow-up (night 2)
  Calculated as sum of Stage 1, 2 and 3 sleep (in minutes and % of total sleep time). A one-way ANCOVA will be computed with baseline non-rapid eye movement sleep (in minutes and % of total sleep time) and minimization factors as covariates, intervention as the independent variable, and follow-up non-rapid eye movement sleep (in minutes and % of total sleep time) as dependent variables.
Change from baseline in rapid eye movement sleep-latency (minutes) at follow-up assessed by polysomnography | Baseline (night 1) and follow-up (night 2)
  Calculated as time between sleep onset and the occurrence of the first REM sleep epoch (minutes). A one-way ANCOVA will be computed with baseline rapid eye movement sleep-latency (minutes) and minimization factors as covariates, intervention as the independent variable, and follow-up rapid eye movement sleep-latency (minutes) as dependent variables.
Change from baseline in stage shift index at follow-up assessed by polysomnography | Baseline (night 1) and follow-up (night 2)
  Calculated as the number of transitions between any wake or sleep stage divided by hours of total sleep time. Lower values represent better outcome. A one-way ANCOVA will be computed with baseline stage shift index and minimization factors as covariates, intervention as the independent variable, and follow-up stage shift index as dependent variables.
Change from baseline in subjective sleep quality at follow-up assessed by self-rated questionnaire 'revised Schlaffragebogen A' | Baseline (night 1) and follow-up (night 2)
  Five factors are calculated from 'revised Schlaffragebogen A': sleep quality, recuperation after sleep, calmness prior to sleep, exhaustion prior to sleep, and psychosomatic symptoms during sleep. Values range from 1 to 5. Higher values indicate better outcome in the first three subscales. Lower values indicate better outcome in the last two subscales. A one-way ANCOVA will be computed with baseline values and minimization factors as covariates, intervention as the independent variable, and follow-up value as dependent variables.
Change from baseline in subjective pre-sleep arousal at follow-up assessed by self-rated questionnaire 'Pre-Sleep Arousal Scale' | Baseline (night 1) and follow-up (night 2)
  Two factors are calculated from 'Pre-Sleep Arousal Scale': cognitive arousal (range: 7-35) and somatic arousal (range: 8-40). Lower values indicate better outcome in both scales. A one-way ANCOVA will be computed with baseline values and minimization factors as covariates, intervention as the independent variable, and follow-up value as dependent variables.
Change from baseline in pre-sleep autonomic modulation at follow-up | Baseline (night 1) and follow-up (night 2)
  Assessed through short-term (5 minutes as of lights off) heart rate variability measured by ECG (modified lead II). Heart rate variability will be assessed by time-domain (Root Mean Square of successive differences of normal-to-normal intervals (RMSSD) and standard deviation of normal-to-normal intervals (SDNN)) as well as frequency domain (total power (TP), low frequency power (LF), high frequency power (HF), and ratio of LF-to-HF power (LF/HF)). A one-way ANCOVA will be computed with baseline heart rate variability indices and minimization factors as covariates, intervention as the independent variable, and follow-up heart rate variability indices as the dependent variable.
Change from baseline in nocturnal autonomic modulation at follow up | Baseline (night 1) and follow-up (night 2)
  Assessed by heart rate variability through a 6-hour period as of sleep onset, measured by ECG (modified lead II). Heart rate variability will be assessed by time-domain (Root Mean Square of successive differences of normal-to-normal intervals (RMSSD) and standard deviation of normal-to-normal intervals (SDNN)) as well as frequency domain (total power (TP), low frequency power (LF), high frequency power (HF), and ratio of LF-to-HF power (LF/HF)). The 6-hour period is split into six hourly segments for analysis. Hourly segments of nocturnal HRV will be analyzed using a linear mixed model with subject as random effect, adjusting for baseline and minimization factors.
Change from baseline in post-sleep autonomic modulation at follow-up | Baseline (night 1) and follow-up (night 2)
  Assessed through short-term (5 minutes as of last awakening) heart rate variability measured by ECG (modified lead II). Heart rate variability will be assessed by time-domain (Root Mean Square of successive differences of normal-to-normal intervals (RMSSD) and standard deviation of normal-to-normal intervals (SDNN)) as well as frequency domain (total power (TP), low frequency power (LF), high frequency power (HF), and ratio of LF-to-HF power (LF/HF)). A one-way ANCOVA will be computed with baseline heart rate variability indices and minimization factors as covariates, intervention as the independent variable, and follow-up heart rate variability indices as the dependent variable.
Change from baseline in nocturnal mean arterial pressure at follow-up assessed by pulse transit time (ECG, modified lead II; fingertip photoplethysmogram, single initial calibration measurement) | Baseline (night 1) and follow-up (night 2)
  Mean arterial pressure is calculated from systolic and diastolic blood pressures as follows: [(0.33 * systolic pressure) + (0.66 * diastolic pressure)]. Mean arterial pressure will be reported separately for total sleep time, non-rapid eye movement sleep, and rapid eye movement sleep. A one-way ANCOVA will be computed with baseline mean arterial pressure and minimization factors as covariates, intervention as the independent variable, and follow-up mean arterial pressure as the dependent variable.
State sleepiness assessed by self-rated questionnaire 'Stanford Sleepiness Scale' (SSS) | Day 5 (i.e. day after night 2): at 08:00 am, 12 noon, 04:00 pm, and 08:00 pm
  This is a single item questionnaire on a 7-point scale (1-7). Higher values indicate worse outcome.
Difference in adverse events between exercise and control group | Immediately after termination of exercise intervention or control condition and after awakening from follow-up (night 2)
  Adverse events will be explicitly assessed through a questionnaire. Patients will be asked whether they experienced adverse effects on a five point Likert scale (not at all, very) using the following categories: Pain (if yes, location), dizziness, cardiovascular symptoms (e.g. angina symptoms, cyanosis, pallor), respiratory symptoms (e.g. wheezing), nausea, falls (yes or no), other (to be described).

OTHER OUTCOMES:
Mood assessed by self-rating questionnaire 'Befindlichkeitsskala' (BFS) | Immediately before and at the end of the control condition as well as the exercise intervention.
  Eight subscales are calculated from the 'Befindlichkeitsskala' (BFS): activity, elation, contemplation, calmness, fatigue, depression, anger, and excitement. Values of all subscale range from 1 to 5. Higher scores on the subscale depression indicate worse outcome. Higher scores on the other subscales cannot a priori be judged as representing better or worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Brupbacher, MSc, Principal Investigator — Oberwaid AG; Hildburg Hildburg, MD, Principal Investigator — Oberwaid AG
Locations (1):
- Oberwaid Ag, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
De-identified (i.e. coded) individual participant data that underlie the results of published articles, including data dictionaries, will be available upon request under the creative commons license CC-BY. Requests will only be granted for use in individual participant data meta-analysis which has been approved by an independent review committee. Exceptions to these rules are reserved within the context of peer-reviewed publications, provided that data integrity remains intact. Data will be provided upon request immediately after publication of peer-reviewed articles with no end date. Requests should be sent to the e-mail address detailed in the Dataverse repository https://doi.org/10.7910/DVN/WASN36.
Supporting Information: Study Protocol
URL: https://doi.org/10.7910/DVN/WASN36

REFERENCES:
- [Derived] Brupbacher G, Zander-Schellenberg T, Straus D, Porschke H, Infanger D, Gerber M, von Kanel R, Schmidt-Trucksass A. The acute effects of aerobic exercise on sleep in patients with unipolar depression: a randomized controlled trial. Sleep. 2021 Nov 12;44(11):zsab177. doi: 10.1093/sleep/zsab177. PMID 34255075
- [Derived] Brupbacher G, Straus D, Porschke H, Zander-Schellenberg T, Gerber M, von Kanel R, Schmidt-Trucksass A. The acute effects of aerobic exercise on sleep in patients with depression: study protocol for a randomized controlled trial. Trials. 2019 Jun 13;20(1):352. doi: 10.1186/s13063-019-3415-3. PMID 31196147
- Available data/document: Individual Participant Data Set — https://doi.org/10.7910/DVN/WASN36